CLINICAL TRIAL: NCT02811666
Title: Impact of Preoperative Sarcopenia on Morbidity and Mortality in Patients Operated on From Digestive Cancers
Acronym: A15-10
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PA16063
Record Dates: First submitted 2016-06-17; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Sarcopenia; Malnutrition; Pancreatic Cancer; Liver Cancer
MeSH Terms: conditions — Sarcopenia; Malnutrition; Pancreatic Neoplasms; Liver Neoplasms

ARMS (1):
- Patients operated for liver or pancreas cancer (Experimental)
  Interventions: Device: Assessment of sarcopenia by CT-Scan; Device: hand gauge

INTERVENTIONS:
Device: Assessment of sarcopenia by CT-Scan
Device: hand gauge

SUMMARY:
Sarcopenia (loss of muscle mass and function) can be observed at any age and results of multiple factors (age, activity, inflammatory factors, nutritional status...). It deeply impacts the physical performance and the basal metabolism, and induces cardiovascular disorders, dyslipidemia, and diabetes. Sarcopenia appears like an independent factor decreasing the quality of life, exacerbating the toxicity of chemotherapy and increasing mortality for gastrointestinal cancer. However, few studies have demonstrated his impact on postoperative course in digestive oncology. The search for sarcopenia, complementary nutritional status, is now a source of great interest with 62 ongoing projects in the United States.

The first objective of this study is to evaluate the impact of preoperative sarcopenia on 30-days morbidity and mortality of patients operated on from poor prognosis gastrointestinal cancer (liver and pancreas). The second objective is to evaluate the impact of preoperative sarcopenia on the long term outcomes (12 months) on the same patients.

DETAILED DESCRIPTION:
In this interventional, intent-to-treat, single-center cohort, prospective study, sarcopenia will be evaluated by the decrease in muscle surface (assessed by CT-Scan) associated with a decrease in muscle strength (assessed by hand gauge). Preoperative evaluation will also include nutritional status by physical examination and laboratory tests, and many nutritional questionnaires. The same data (including sarcopenia, laboratory tests and nutritional evaluation) will be collected at 7 days, 30 days and 12 months, as well as the morbidity and mortality. Statistical tests might evaluate if sarcopenia may be an independent factor of morbidity and mortality among these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in the our digestive surgery department during the inclusion phase for the surgical curative treatment of liver (primary or secondary) and pancreatic cancer
* Patients over 18 years
* Patients who agreed to participate in the study
* The patients insured by French health care

Exclusion Criteria:

* Patients treated by radio-frequency
* Patients operated for extrahepatic cholangiocarcinoma , cancer of the papilla of Vater or the gall-bladder
* Patients with primary peritoneal cancer
* Patients with palliative surgery without resection
* Patients protected by law
* Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
muscle surface using CT-Scan | up to12th month postoperatively
muscle strength using a hand gauge | up to12th month postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France